CLINICAL TRIAL: NCT01342406
Title: Effects of Selective Laser Trabeculoplasty on Aqueous Humor Dynamics
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0191-10-FB
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will compare aqueous humor dynamics in adults with primary open angle glaucoma that receive Selective Laser Trabeculoplasty (SLT).

DETAILED DESCRIPTION:
Describe the background of the study. Include a critical evaluation of existing knowledge, and specifically identify the information gaps that the project is intended to fill.

Laser trabeculoplasty is currently a well established treatment option for lowering the intraocular pressure in the management of open angle glaucoma1,2. The procedure involves placement of laser spots over the trabecular meshwork, possibly through a variety of laser types. Argon laser trabeculoplasty (ALT) has been the most widely utilized option for laser trabeculoplasty over the past few decades. Since its availability approximately a decade ago, Selective Laser Trabeculoplasty (SLT) is currently an additional option for doing laser trabeculoplasty. 3,4. Current evidence suggests that SLT achieves its interocular pressure (IOP) lowering effect without thermal damage to the trabecular meshwork5. The IOP lowering effect of SLT has been shown to be comparable to ALT over the long term6.

In physiological terms, ALT has been shown to lower the IOP primarily by increasing the conventional outflow facility7. There are two putative mechanisms by which this may be facilitated8. Thermal coagulation and shrinkage by ALT may mechanically open up the adjacent trabecular meshwork and Schlemm's canal. Alternatively the delivery of laser energy may trigger biological processes and activation of matrix metalloproteinases in the microenvironment of trabecular meshwork that lead to a remodeling of tissues resulting in improved outflow facility. ALT uses argon or another thermal laser to photocoagulate tissues around the trabecular meshwork. The settings vary depending on the tissue response and pigmentation. Most clinicians use 600-1500mW, 50-100 spots, 50 micron spot size and 0.1 sec duration.

Also, there is limited data on fluorophotometric and tonographic studies on ALT and none on SLT to the best of our knowledge. All available reference known to the investigators have been included in the list of references.

The effect of SLT on the aqueous humor dynamics is currently unknown. Given the lack of demonstrable thermal damage on histopathologic examination5, it is unlikely that the effects of SLT could be mechanically mediated. There has been some suggestion of a potential interaction of IOP lowering effect when prostaglandins and SLT are used together9,10. This suggests that there could be a possible sharing of mechanisms between SLT and prostaglandins. The IOP lowering effect of SLT may be mediated in part by effects on uveoscleral pathways in addition to the trabecular outflow pathway. This study will determine the changes in aqueous humor dynamics produced by SLT that lead to its IOP lowering effect. SLT is a Q switched frequency doubled Nd:YAG laser. The duration is 3 nanoseconds and spot size 500 microns. Power varies from 0.5-1.5 mJ and total number of spots can be between 50-over 100. The mechanism of action may be disruption of melanosomes, but this has not been unequivocally proven yet.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age and older
* Eye consideration for SLT (intraocular pressure above target with current medications, intolerance/allergy to topical medications, patient preference as primary treatment)
* Open angles on gonioscopy

Exclusion Criteria:

* Any previous surgical or laser procedures
* Secondary glaucoma including pigmentary, exfoliative, uveitic, and traumatic glaucomas
* Corneal opacities interfering with adequate fluorophotometry
* Any active ocular infection within the past 2 months
* Any corneal pathology increasing the likelihood of corneal abrasions
* Inability to safely washout medications prior to laser treatment
* Allergies to fluorescein, timolol, dorzolamide, or sulfa
* Excessive (3+) trabecular meshwork pigmentation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with open angle glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2013-11-01 (Actual); Study Completion 2013-11-01 (Actual)

PRIMARY OUTCOMES:
Changes in intraocular pressure (IOP) after Selective Laser Trabeculoplasty (SLT) and changes in outflow facility | 3 years
  This study will compare aqueous humor dynamics (intraocular pressure) in adults with primary open angle glaucoma that receive Selective Laser Trabeculoplasty (SLT).

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Gulati, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Department of Ophthalmology, Omaha, Nebraska, United States